CLINICAL TRIAL: NCT05678972
Title: Pause and Breathe: Online Self-Help Mindfulness-Based Intervention: Investigation of Its Efficacy and Mechanism of Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Winnie W.S. MAK, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBRE-22-0350
Record Dates: First submitted 2023-01-09; First posted 2023-01-10 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Mindfulness
Keywords: Mindfulness; Non-attachment; Internet-based mindfulness-based intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness group (Experimental): Participants in the mindfulness group will be expected to complete a self-help online mindfulness-based intervention, delivered over a 4-week period via an e-learning mental health platform. They will be assessed at three different time points: (1) before the intervention (pre-test assessment), (2) right after the 4-week intervention (post-test assessment), and (3) four weeks after the intervention (follow-up assessment).
  Interventions: Other: Self-help online mindfulness-based intervention
- Waitlist control group (No Intervention): The participants in waitlist control group will be offered access to the online mindfulness course after the study has ended.

INTERVENTIONS:
Other: Self-help online mindfulness-based intervention — This self-help online mindfulness-based intervention is comprised of four weekly modules on education about mindfulness, guided meditations (e.g., mindful breathing, mindful eating, mindful walking, body scan, acceptance, choiceless awareness and disengaging from thoughts exercise), and guidance on using informal mindfulness skills in day-to-day life. Readings, audio and videos are included to explain the concept of mindfulness and overcome common difficulties associated with mindfulness practice.
  Participants will be asked to meditate daily and complete a daily log on their mindfulness practice during this 8-week period.
  Arms: Mindfulness group

SUMMARY:
The current study aims to evaluate the effectiveness of a 4-week self-help online mindfulness-based intervention on mental and physical well-being in comparison to the waitlist control group. This study can provide support to the utility of self-help online mindfulness-based intervention, which may advance our understanding of the causal pathways between mindfulness-based intervention and well-being and guide future research. It is hypothesized that participants in the experimental condition will show better mental well-being, physical well-being, and better improvement in mindfulness and related attributes compared with participants in the control condition.

Upon completing the screening and pre-evaluation questionnaire, participants will be randomly assigned to either mindfulness group or waitlist control group. They will complete three sets of questionnaires in total which will be administered before the intervention (pre-test assessment), right after the 4-week intervention (post-test assessment), and four weeks after the intervention (follow-up assessment), respectively. In the experimental group, participants in the mindfulness group will engage in a 4-week online mindfulness course. The self-help online mindfulness course includes education about mindfulness, guided meditations (e.g., mindful breathing, mindful eating, mindful walking, body scan, acceptance, choiceless awareness and disengaging from thoughts exercise), and guidance on using informal mindfulness skills in day-to-day life. Readings, audio and videos are included to explain the concept of mindfulness and overcome common difficulties associated with mindfulness practice. In the waitlist control group, participants are to refrain from access the online course until they finished the follow-up questionnaire. All participants will be able to access the materials in an online platform after they have completed the research.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over age 18
* Have access to computer and mobile phone (since this is an internet-based study)
* Have ability to read and comprehend Cantonese

Exclusion Criteria:

* Completion of mindfulness-related program/research in the past 3 months
* Have regular mindfulness practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 939 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Mindfulness and discernment | at baseline
  Mindfulness and discernment will be assessed using the Mindfulness-Discernment Scale. Ten items capture participants' levels of mindfulness and fourteen items reflect participants' levels of discernment. Items are rated on a scale ranging from 1 (Never) to 6 (Always).
Mindfulness and discernment | 4th week
  Mindfulness and discernment will be assessed using the Mindfulness-Discernment Scale. Ten items capture participants' levels of mindfulness and fourteen items reflect participants' levels of discernment. Items are rated on a scale ranging from 1 (Never) to 6 (Always).
Mindfulness and discernment | 8th week
  Mindfulness and discernment will be assessed using the Mindfulness-Discernment Scale. Ten items capture participants' levels of mindfulness and fourteen items reflect participants' levels of discernment. Items are rated on a scale ranging from 1 (Never) to 6 (Always).

SECONDARY OUTCOMES:
Mental Well-being | at baseline, 4th, and 8th week
  The Warwick Edinburgh Mental Well-being Scale (Tennant et al, 2007). The WEMWBS is a measure of mental well-being focusing entirely on positive aspects of mental health. It is a 7-item measure, using a 5-point Likert scale from 1 (none of the time) to 5 (all of the time).
  The Warwick Edinburgh Mental Well-being Scale (Tennant et al, 2007) WEMWBS is a measure of mental well-being focusing entirely on positive aspects of mental health. It is a 7-item measure, using a 5-point Likert scale from 1 (none of the time) to 5 (all of the time).
Non-attachment | at baseline, 4th, and 8th week
  The Nonattachment Scale-Short Form (Chio, Lai, & Mak, 2018) was used to measure nonattachment. Participants rated the items from 1 (disagree strongly) to 6 (agree strongly). Excellent internal consistency was demonstrated in the previous studies.
Psychological distress | at baseline, 4th, and 8th week
  Psychological distress will be measured by the 6-item Kessler Psychological Distress Scale, which is a well-established measure on psychological distress that asks about a person's emotional state from 0 (none of the time) to 4 (all of the time).
Physical well-being | at baseline, 4th, and 8th week
  Visual Analogue Scale-Pain (VAS-P), Visual Analogue Scale-Energy (VAS-E), and Sleep disturbance subscale of the Medical Outcomes Study Sleep Measure (MOS-Sleep) will be used to assess participants' physical well-being. Participants will rate items related to their subjective energy level , pain and sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sun Y, Luk TT, Wang MP, Shen C, Ho SY, Viswanath K, Chan SSC, Lam TH. The reliability and validity of the Chinese Short Warwick-Edinburgh Mental Well-being Scale in the general population of Hong Kong. Qual Life Res. 2019 Oct;28(10):2813-2820. doi: 10.1007/s11136-019-02218-5. Epub 2019 May 29. PMID 31144205
- [Background] Staples LG, Dear BF, Gandy M, Fogliati V, Fogliati R, Karin E, Nielssen O, Titov N. Psychometric properties and clinical utility of brief measures of depression, anxiety, and general distress: The PHQ-2, GAD-2, and K-6. Gen Hosp Psychiatry. 2019 Jan-Feb;56:13-18. doi: 10.1016/j.genhosppsych.2018.11.003. Epub 2018 Nov 22. PMID 30508772
- [Background] Tsoi EWS, Tong ACY, Mak WWS. Nonattachment at Work on Well-being Among Working Adults in Hong Kong. Mindfulness (N Y). 2022;13(10):2461-2472. doi: 10.1007/s12671-022-01971-y. Epub 2022 Sep 5. PMID 36089936
- [Background] Schneider D, Appleton L. A reason for visit classification system for ambulatory care. Med Rec News. 1976 Oct;47(5):59-66, 68. No abstract available. PMID 1028884
- [Background] Joyce CR, Zutshi DW, Hrubes V, Mason RM. Comparison of fixed interval and visual analogue scales for rating chronic pain. Eur J Clin Pharmacol. 1975 Aug 14;8(6):415-20. doi: 10.1007/BF00562315. PMID 1233242
- [Background] Folstein MF, Luria R. Reliability, validity, and clinical application of the Visual Analogue Mood Scale. Psychol Med. 1973 Nov;3(4):479-86. doi: 10.1017/s0033291700054283. No abstract available. PMID 4762224
- [Background] O'Connor PJ. Mental energy: Assessing the mood dimension. Nutr Rev. 2006 Jul;64(7 Pt 2):S7-9. doi: 10.1111/j.1753-4887.2006.tb00256.x. PMID 16910215
- [Background] Sahdra BK, Shaver PR, Brown KW. A scale to measure nonattachment: a Buddhist complement to Western research on attachment and adaptive functioning. J Pers Assess. 2010 Mar;92(2):116-27. doi: 10.1080/00223890903425960. PMID 20155561